CLINICAL TRIAL: NCT02071719
Title: Prediction of Response to Kinase Inhibitors Based on Protein Phosphorylation Profiles in Tumor Tissue From Advanced Renal Cell Cancer Patients
Status: Terminated | Type: Observational
Sponsor: M. Labots (Other)
Responsible Party: Sponsor-Investigator, M. Labots, Medical Oncologist, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Other Study IDs: 2012/109
Record Dates: First submitted 2012-12-11; First posted 2014-02-26 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Sunitinib
- Sorafenib
- Everolimus
- Pazopanib
- Axitinib

SUMMARY:
The rapid development of agents blocking kinases has established the use of molecularly targeted therapy as the preferred treatment approach for patients with metastatic renal cell cancer (RCC). Five kinase inhibitors (sunitinib, everolimus, temsirolimus, sorafenib and pazopanib) are now approved for clinical use. Response rates differ among these agents, importantly depending on line of treatment. In first-line treatment sunitinib results in 47% objective response rates, where in second-line after cytokines 34% responds. Thus far, it is unclear which patient with advanced renal cell cancer will respond to targeted therapy. In order to select patients for targeted therapies, several profiling approaches have been explored but to date no adequate and reliable test is available. It is assumed that responses to targeted agents depend on specific receptor and protein signalling activities in tumor tissues. Therefore, we propose that protein phosphorylation profiling with phosphoproteomics may be a potential clinical diagnostic tool to predict for tumor response to targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced (unresectable and/or metastatic) renal cell cancer.
* Patients who will start treatment with sunitinib, pazopanib, sorafenib, axitinib or everolimus.
* At least one tumor lesion should be accessible for biopsy. Bone metastases are excluded as possible biopsy site.
* Age >- 18 years.
* Patients must have at least one measurable lesion. Lesions must be evaluated by CT-scan or MRI according to Response Evaluation Criteria in Solid Tumors (RECIST).
* WHO performance status 0 - 2
* Able to provide written informed consent

Exclusion Criteria:

* Clinical findings associated with an unacceptably high tumor biopsy risk, according to the judgement of the investigator.
* Radiotherapy on target lesions during study or within 4 weeks of the start of drug.
* Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with renal cell cancer
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-04; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Response to treatment | Follow up once every 4 months until disease progression or death of the patient
Progression Free Survival | once every 4 months until disease progression or death of the patient
  To determine the relation between tumor tissue phosphoproteomic profiles and progression-free survival (PFS) in patients with advanced RCC

SECONDARY OUTCOMES:
PamChip kinase activity profiling and PFS | Sample collection at inclusion is mandatory (1). Collection after 2-4 weeks of treatment (2) and upon progression (3) are optional
genome-wide mutational profiles by Massively Parallel Sequencing (MPS) | Sample collection at inclusion is mandatory (1). Collection after 2-4 weeks of treatment (2) and upon progression (3) are optional
serum proteomic profiles | Sample collection at inclusion is mandatory (1). Collection after 2-4 weeks of treatment (2) and upon progression (3) are optional
the value of the frequency and phenotype of immunoregulatory cells in blood and tumor tissue | Sample collection at inclusion is mandatory (1). Collection after 2-4 weeks of treatment (2) and upon progression (3) are optional
genetic polymorphisms and pharmacokinetic parameters | Sample collection at inclusion is mandatory (1). Collection after 2-4 weeks of treatment (2) and upon progression (3) are optional
tumor exosomes from urine and serum | Sample collection at inclusion is mandatory (1). Collection after 2-4 weeks of treatment (2) and upon progression (3) are optional

CONTACTS AND LOCATIONS:
Locations (1):
- VU Medical Center, Amsterdam, North Holland, Netherlands